CLINICAL TRIAL: NCT02513524
Title: The Prevalence of Pseudo-resistant Hypertension Using the Direct Observed Therapy Test: A Prospective Observational Study
Brief Title: Prevalence of Resistant Hypertension With DOT
Acronym: DOT
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 4096
Record Dates: First submitted 2015-07-23; First posted 2015-07-31 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Hypertension
Keywords: hypertension; adherence; resistant hypertension; blood pressure; non-adherence
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Direct Observed Therapy test: Patients with resistant hypertension (as defined in the eligibility criteria) will be enrolled. They will all have undergone 24 hour ambulatory blood pressure monitoring (ABPM) before enrollment. As part of the study, the subjects will undergo direct observed therapy testing, followed by another 24 hour ABPM, which will be repeated at 1 month.
  Interventions: Procedure: Direct Observed Therapy test

INTERVENTIONS:
Procedure: Direct Observed Therapy test — There is one group only, all of whom will undergo direct observed therapy testing

SUMMARY:
High blood pressure is a risk factor for bad clinical events, such as heart failure, stroke, kidney failure and death. This risk is much higher in those with 'resistant' hypertension, in whom the blood pressure remains high despite more than 3 blood pressure medicines. Current estimates of the proportion of individuals with resistant hypertension may be an overestimate, since some of them are not actually adherent (i.e. not taking the medicines they are prescribed). Methods to detect non-adherence, such as asking the patient, counting pills, and getting records from pharmacy are not fool proof. Direct observed therapy (where patients are administered medicines under observation by a health care personnel) is quite useful to diagnose this, and is the standard of care in the Renal Hypertension Clinic, before more tests and interventions (such as CT scans, renal angiogram) are performed.

In this study, the investigators will measure the proportion of patients with resistant hypertension who are non-adherent based on direct observed therapy, and follow them up to examine the impact of this diagnosis.

DETAILED DESCRIPTION:
This is a prospective, observational study.

Patients fitting inclusion and exclusion criteria, after informed consent, will undergo the direct observed therapy test in the hypertension unit (this is usual care in the unit, which they will undergo even if they are not part of the study).

The Direct Observation Therapy (DOT) Test includes the following components:

1. Administer and observe ingestion of usual morning antihypertensive medications.
2. Monitor BP every 30 minutes, using 5 readings of an automated oscillometric BP device ( BP-TRU), until plateau affect achieved, defined as 3 consecutive cycles of BP readings declining by less than 10 mmHg per cycle).
3. Registered Nurse (RN) repeats standing BP prior to initiation of 24 hour Ambulatory Blood Pressure Monitoring(ABPM).
4. RN initiates 24 hour ABPM

In addition, participants will undergo an additional 24-hour ABPM test 1 month after the DOT test is undertaken.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Confirmed resistant hypertension defined as daytime BP readings above 135/85 mmHg (confirmed by 24-hour ABPM results) using 3 or more BP lowering drugs
3. Adherence to medications confirmed by patient, and by hypertension clinic on basis of pharmacy filling record

Exclusion Criteria:

1. Pregnant patients
2. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients with resistant hypertension referred to a tertiary care hypertension clinic.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of true resistant hypertension | 1 week
  The proportion of patients who continue to have resistant hypertension after administration of direct observed therapy, on the basis of the 24 hour ambulatory testing

SECONDARY OUTCOMES:
Prevalence of resistant hypertension at 1 month | 1 month
  The proportion of patients who continue to have resistant hypertension at one month, on the basis of the 24 hour ambulatory testing

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Ruzicka, MD PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada